CLINICAL TRIAL: NCT02749292
Title: Maintenance of ANCA Vasculitis Remission by Intermittent Rituximab Dosing Based on B-cell Reconstitution vs a Serologic ANCA Flare
Brief Title: Maintenance of ANCA Vasculitis Remission by Intermittent Rituximab Dosing
Acronym: MAINTANCAVAS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the coronavirus disease 2019 (COVID-19) pandemic and the deleterious impact of rituximab on vaccination efficacy, the trial was concluded before reaching the target enrollment of 200.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John L Niles, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015P002541
Record Dates: First submitted 2016-03-01; First posted 2016-04-22 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis
Keywords: rituximab; maintenance; remission
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B cell reconstitution (Active Comparator): Subjects will not receive their regularly-scheduled every-six-month dose of rituximab and will instead receive rituximab 1000 mg IV x 1 dose once peripheral B cells return ( ≥ 10 B cells/mm3). This cycle will then re-start. Subjects will be seen in clinic every three months. Patients will continue to be dosed with rituximab each time the B cell count rises to 10 cells/mm3. In the unique scenario that the B cells are detectable, but less than the threshold of 10 cells/mm3, subjects will be asked to return in 6 weeks for repeat B cell testing.
  Interventions: Drug: Rituximab
- Serologic ANCA flare (Active Comparator): Subjects will not receive regularly scheduled every six-month doses of rituximab (1000mg IV) and will instead be seen in clinic for ANCA titer monitoring every 3 months. Re-dosing will occur upon a significant ANCA titer increase. For MPO, a significant rise will be defined as a 5-fold rise in ANCA titer and a level greater than 4 times the cutoff value for the assay. For PR3, a significant rise will be defined as a 4-fold rise in ANCA titer to a level at least twofold above the cutoff for the assay. Subjects who sustain a significant increase in ANCA titer will receive rituximab 1000mg IV x 2 doses, spaced ~2-3 weeks apart. If the ANCA titer remains two-fold above baseline and above a specified threshold (the cutoff value of the assay for PR3 and 4 times the cutoff value for MPO) , subjects will continue to receive rituximab 1000mg IV every 6 months for a maximum of 2 doses, at which time a new baseline ANCA titer will be established and the cycle will re-start.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — re-dosing dependent on interventional arm parameter.
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to determine the best management strategy to maintain remission in patients with ANCA vasculitis who have been treated with rituximab induced B cell depletion for at least two years. This study will compare intermittent B Cell depletion upon B cell return or intermittent B cell depletion upon serologic relapse.

DETAILED DESCRIPTION:
Anti-neutrophil cytoplasmic autoantibody (ANCA) vasculitis is a systemic autoimmune disease characterized by small vessel inflammation caused by pathogenic autoantibodies directed against proteinase 3 (PR3) or myeloperoxidase (MPO). Immunosuppressive therapy can result in remission; however, many patients relapse, which results in additional injury.

Rituximab, a humanized murine monoclonal antibody directed against CD20 located on the surface of B-lymphocytes (B cells), is effective in depleting B cells. The RAVE and RITUXVAS trials have shown efficacy of rituximab with steroids for induction of remission in ANCA vasculitis, similar to cyclophosphamide and steroids. Rituximab is now FDA-approved for induction of remission therapy in ANCA vasculitis. The utility of anti-B-cell therapy for early induction of remission in ANCA vasculitis is not surprising given that ANCA are pathogenic in vitro and in vivo. It is clear that remission in many patients is not sustained with a single induction course of rituximab, and relapses often occur after B cell re-population suggesting that scheduled, serial dosing of rituximab could result in sustained remissions.

Despite yielding promising outcomes, rituximab is also associated with a number of adverse events including infectious complications and late onset of neutropenia5, 15. Furthermore, the complications of continuous B cell depletion for extended durations are unknown. One of the major goals in the field is to utilize prolonged B cell depletion only in the subpopulation of patients where the risk of disease relapse outweighs the risk of treatment-related adverse events.

A rise in ANCA titers and reconstitution of B cells are promising biomarkers of impending disease relapse following treatment with rituximab4-6

A prospective and longitudinal clinical trial is needed to determine the ideal treatment strategy for long-term maintenance of remission. We propose to compare intermittent rituximab dosing based on B cell return and a serologic ANCA flare

The study design is an open-label, single center, randomized and two-arm controlled trial to evaluate the optimal maintenance of remission strategy that provides the best relapse-free survival in patients with ANCA vasculitis as determined by relapse-free remission at 18, 24 and 36 months from enrollment. The investigators are looking to enroll and randomize 200 subjects with ANCA vasculitis on rituximab-induced continuous B cell depletion for a minimum of two years to one of two arms as follows:

1. Intermittent B cell depletion with rituximab re-dosing upon B cell return: Subjects will not receive their regularly-scheduled every-six-month dose of rituximab and will instead receive rituximab 1000 mg IV x 1 dose (spaced 2-3 weeks apart) once peripheral B cells return ( ≥ 10 B cells/mm3). This cycle will then re-start. Subjects will be seen in clinic every three months. Patients will continue to be dosed with rituximab each time the B cell count rises to 10 cells/mm3. In the unique scenario that the B cells are detectable, but less than the threshold of 10 cells/mm3, subjects will be asked to return in 6 weeks for repeat B cell testing.
2. Hold continuous dosing with rituximab with re-dosing upon a significant ANCA titer increase: For MPO, a significant increase will be defined as a 5-fold rise in ANCA titer and a level greater than 4 times the cutoff value for the assay. For PR3, a significant rise will be defined as a 4-fold rise in ANCA titer to a level at least twofold above the cutoff for the assay. Subjects will not receive regularly scheduled every six-month doses of rituximab and will instead be seen in clinic to have their ANCA titer monitored every three months. Subjects who sustain a significant increase in ANCA titer will receive rituximab 1000mg IV x 2 doses, ~2-3 weeks apart. If the ANCA titer remains two-fold above baseline and above a specified threshold (the cutoff value of the assay for PR3 and 4 times the cutoff value for MPO) , subjects will continue to receive rituximab 1000mg IV every 6 months for a maximum of 2 doses, at which time a new baseline ANCA titer will be established and the cycle will re-start.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be able and willing to give written informed consent and comply with the requirements of the study protocol.
2. Diagnosis: ANCA vasculitis as defined by a positive MPO- and/or PR3-ANCA test together with clinical features characteristic of ANCA-positive diseases as detailed in the 2012 Chapel Hill Consensus Conference Definitions(18).
3. eGFR ≥ 73 cc/min/1.73m2
4. Age: 18-82 years old
5. Treated with rituximab-induced continuous B cell depletion at regularly scheduled interval with a goal of undetectable B cells for at least 24 months
6. In sustained remission (defined by a modified BVAS-WG=0 AND a prednisone dose of ≤ 7.5 mg) for at least 12 months.
7. Undetectable (<10mm3) B cells (quantified by CD20+ number) on day 0
8. Urine Hcg negative for women of child bearing potential and not planning to become pregnant for at least 12 months from enrollment and at least 12 months after any study related rituximab dose
9. Judged to be otherwise healthy by the Investigator, based on medical history and physical examination (no known active disease process for which life expectancy is less than 36 months)

Exclusion Criteria:

1. Secondary Disease: disease suspected to be induced by levamisole-adulterated cocaine
2. All transplanted patients
3. Treatment: additional immunosuppressive agents other than rituximab and/or total daily prednisone dose ≥ 7.5 milligrams
4. Hypogammaglobulinemia: IgG level < 300 mg/dL
5. Terminal cancer or other primary illness with life expectancy of less than 36 months
6. Active anti-GBM disease and other known autoimmune disease for which the need for additional immunosuppression is likely
7. Pregnancy or breastfeeding

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2016-06; Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John L Niles, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jennette JC, Falk RJ, Gasim AH. Pathogenesis of antineutrophil cytoplasmic autoantibody vasculitis. Curr Opin Nephrol Hypertens. 2011 May;20(3):263-70. doi: 10.1097/MNH.0b013e3283456731. PMID 21422922
- [Background] Jones RB, Tervaert JW, Hauser T, Luqmani R, Morgan MD, Peh CA, Savage CO, Segelmark M, Tesar V, van Paassen P, Walsh D, Walsh M, Westman K, Jayne DR; European Vasculitis Study Group. Rituximab versus cyclophosphamide in ANCA-associated renal vasculitis. N Engl J Med. 2010 Jul 15;363(3):211-20. doi: 10.1056/NEJMoa0909169. PMID 20647198
- [Background] Stone JH, Merkel PA, Spiera R, Seo P, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Turkiewicz A, Tchao NK, Webber L, Ding L, Sejismundo LP, Mieras K, Weitzenkamp D, Ikle D, Seyfert-Margolis V, Mueller M, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh KA, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Specks U; RAVE-ITN Research Group. Rituximab versus cyclophosphamide for ANCA-associated vasculitis. N Engl J Med. 2010 Jul 15;363(3):221-32. doi: 10.1056/NEJMoa0909905. PMID 20647199
- [Background] Jayne D, Rasmussen N, Andrassy K, Bacon P, Tervaert JW, Dadoniene J, Ekstrand A, Gaskin G, Gregorini G, de Groot K, Gross W, Hagen EC, Mirapeix E, Pettersson E, Siegert C, Sinico A, Tesar V, Westman K, Pusey C; European Vasculitis Study Group. A randomized trial of maintenance therapy for vasculitis associated with antineutrophil cytoplasmic autoantibodies. N Engl J Med. 2003 Jul 3;349(1):36-44. doi: 10.1056/NEJMoa020286. PMID 12840090
- [Background] Specks U, Merkel PA, Seo P, Spiera R, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Fessler BJ, Ding L, Viviano L, Tchao NK, Phippard DJ, Asare AL, Lim N, Ikle D, Jepson B, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh K, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Mueller M, Sejismundo LP, Mieras K, Stone JH; RAVE-ITN Research Group. Efficacy of remission-induction regimens for ANCA-associated vasculitis. N Engl J Med. 2013 Aug 1;369(5):417-27. doi: 10.1056/NEJMoa1213277. PMID 23902481
- [Background] Pendergraft WF 3rd, Cortazar FB, Wenger J, Murphy AP, Rhee EP, Laliberte KA, Niles JL. Long-term maintenance therapy using rituximab-induced continuous B-cell depletion in patients with ANCA vasculitis. Clin J Am Soc Nephrol. 2014 Apr;9(4):736-44. doi: 10.2215/CJN.07340713. Epub 2014 Mar 13. PMID 24626432
- [Background] Guillevin L, Pagnoux C, Karras A, Khouatra C, Aumaitre O, Cohen P, Maurier F, Decaux O, Ninet J, Gobert P, Quemeneur T, Blanchard-Delaunay C, Godmer P, Puechal X, Carron PL, Hatron PY, Limal N, Hamidou M, Ducret M, Daugas E, Papo T, Bonnotte B, Mahr A, Ravaud P, Mouthon L; French Vasculitis Study Group. Rituximab versus azathioprine for maintenance in ANCA-associated vasculitis. N Engl J Med. 2014 Nov 6;371(19):1771-80. doi: 10.1056/NEJMoa1404231. PMID 25372085
- [Background] Han WK, Choi HK, Roth RM, McCluskey RT, Niles JL. Serial ANCA titers: useful tool for prevention of relapses in ANCA-associated vasculitis. Kidney Int. 2003 Mar;63(3):1079-85. doi: 10.1046/j.1523-1755.2003.00821.x. PMID 12631091
- [Background] Alberici F, Smith RM, Jones RB, Roberts DM, Willcocks LC, Chaudhry A, Smith KG, Jayne DR. Long-term follow-up of patients who received repeat-dose rituximab as maintenance therapy for ANCA-associated vasculitis. Rheumatology (Oxford). 2015 Jul;54(7):1153-60. doi: 10.1093/rheumatology/keu452. Epub 2014 Dec 3. PMID 25477054
- [Derived] Zonozi R, Cortazar FB, Jeyabalan A, Sauvage G, Nithagon P, Huizenga NR, Rosenthal JM, Sipilief A, Cosgrove K, Laliberte KA, Rhee EP, Pendergraft WF 3rd, Niles JL. Maintenance of remission of ANCA vasculitis by rituximab based on B cell repopulation versus serological flare: a randomised trial. Ann Rheum Dis. 2024 Feb 15;83(3):351-359. doi: 10.1136/ard-2023-224489. PMID 38123922

RESULTS

PARTICIPANT FLOW:
Groups:
- B Cell Reconstitution: Subjects will not receive their regularly-scheduled every-six-month dose of rituximab (1000mg IV) and will instead receive rituximab 1000 mg IV x 1 dose only once peripheral B cells return ( ≥ 10 B cells/mm3). This cycle will then re-start. Subjects will be seen in clinic every three months. Patients will continue to be dosed with rituximab (1 dose of 1000mg IV) each time the B cell count rises to 10 cells/mm3. In the unique scenario that the B cells are detectable, but less than the threshold of 10 cells/mm3, subjects will be asked to return in 6 weeks for repeat B cell testing.
  Rituximab: re-dosing dependent on interventional arm parameter.
- Serologic ANCA Flare: Subjects will not receive regularly scheduled every six-month doses of rituximab (1000mg IV) and will instead be seen in clinic for ANCA titer monitoring every 3 months. Re-dosing will occur upon a significant ANCA titer increase. For MPO, a significant rise will be defined as a 5-fold rise in ANCA titer and a level greater than 4 times the cutoff value for the assay. For PR3, a significant rise will be defined as a 4-fold rise in ANCA titer to a level at least twofold above the cutoff for the assay. Subjects who sustain a significant increase in ANCA titer will receive rituximab 1000mg IV x 2 doses, spaced ~2-3 weeks apart. If the ANCA titer remains two-fold above baseline and above a specified threshold (the cutoff value of the assay for PR3 and 4 times the cutoff value for MPO) , subjects will continue to receive rituximab 1000mg IV every 6 months for a maximum of 2 doses, at which time a new baseline ANCA titer will be established and the cycle will re-start. In this arm, rituximab administration is not contingent upon B cell levels but on significant ANCA titer rise as described above. Baseline ANCA titer will be recalculated to an average of the two highest of the last four values if all four are less than the original baseline. Patients in the ANCA arm will move to once yearly CD20 testing after CD20 levels return to normal levels (>90 cells/uL).
Period: Overall Study
Arm/Group | B Cell Reconstitution | Serologic ANCA Flare
Started | 58 | 57
Completed (Subjects who were not withdrawn from the study and reached to common close out of the study.) | 36 | 31
Not Completed | 22 | 26
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Minor relapse, BVAS-WG = 2 | 1 | 7
Not completed — Major relapse without ILD, BVAS-WG ≥ 3 | 2 | 4
Not completed — Major relapse with ILD, BVAS-WG ≥ 3 | 2 | 3
Not completed — Adverse Event | 4 | 1
Not completed — Serious Adverse Event, Related, infection, COVID-19, with death | 2 | 0
Not completed — Serious Adverse Event, Related, infection, COVID-19, without death | 4 | 1
Not completed — Requiring glucocorticoids | 0 | 3
Not completed — Cancer | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B Cell Reconstitution | Serologic ANCA Flare | Total
Number analyzed (Participants) | 58 | 57 | 115
Age, Categorical [Count of Participants; unit: Participants] — Age reported is the age of each participant at the time of enrollment. Only subjects aged 18-82 years old were enrolled in the study (inclusion criteria).
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 36 | 34 | 70
    >=65 years | 22 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] — Age reported are based on age of subjects at time of enrollment. Means reported are the arithmetic means and each of the standard deviations was calculated based on the sample/ group for which it was calculated.
  years | 61 (10) | 62 (12) | 61 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 26 | 56
  Male | 28 | 31 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 58 | 56 | 114
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was self-reported by the participants at the time of enrollment, two participants indicated no to each choice of race available. One other participant put "Other" as their race and so the three participants were counted as "Unknown or not Reported" in this report.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 1 | 3
    White | 55 | 53 | 108
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 58 | 57 | 115
ANCA serotype [Count of Participants; unit: Participants]
  Anti-PR3 | 31 | 31 | 62
  Anti-MPO | 27 | 26 | 53
Continuous Rituximab prior to entry [Count of Participants; unit: Participants]
  Less than 3 years at entry | 29 | 28 | 57
  More than 3 years at entry | 29 | 29 | 58
Induction Regimen- Rituximab and Cyclophosphamide [Count of Participants; unit: Participants]
  Cyclophosphamide | 10 | 12 | 22
  Rituximab | 16 | 13 | 29
  Cyclophosphamide and Rituximab | 32 | 32 | 64
Induction Regimen- Plasma Exchange [Count of Participants; unit: Participants] | 12 | 9 | 21
Clinical manifestations at diagnosis [Count of Participants; unit: Participants] — Number of participants presenting with a specific clinical manifestation of ANCA-associated vasculitis at the time of diagnosis. Clinical manifestations are non-exclusive
  Participants
    Scleritis | 18 | 13 | 31
    Otitis | 17 | 17 | 34
    Sinusitis | 30 | 26 | 56
    Tracheal Stenosis | 2 | 2 | 4
    Pulmonary Hemorrhage | 6 | 13 | 19
    ILD | 2 | 1 | 3
    Renal involvement (including RPGN, required Hemodialysis and HD dependent) | 31 | 30 | 61
    Rapidly Progressive Glomerulonephritis (RPGN) | 20 | 15 | 35
    Required Hemodialysis | 1 | 1 | 2
    HD dependent | 0 | 0 | 0
BVAS/WG at entry [Median (Standard Deviation); unit: units on a scale] — The Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG ) is a form with 34 predefined items grouped into 9 organ systems. The items are clinical features observed in patients with active ANCA vasculitis. Each item has a specified weight of either 3 or 1, depending on whether it reflects major or minor disease activity. The total BVAS/WG score is the weighted sum of individual manifestations that are present and believed to be due to active ANCA vasculitis. Higher scores reflect more active disease. BVAS/WG scores range from 0 to 64.
  units on a scale | 0 (0) | 0 (0) | 0 (0)
VDI at entry [Median (Standard Deviation); unit: units on a scale] — The Vasculitis Damage Index (VDI) is a validated formal assessment tool in ANCA-associated vasculitis clinical trials. The VDI distinguishes vasculitis-induced chronic damage from active inflammation or persistent disease. Each item (disease manifestation) is given a score (of 1) if present for at least 3 months. Neither the cause of damage nor an ongoing activity are taken into consideration. The VDI includes 64 items categorized into 11 groups (by organ system) and the scored items are summed to give a total score ranging from 0 to 64. A higher score means more accrued damage.
  units on a scale | 1 (1) | 1 (1) | 1 (1)
Creatinine at entry [Median (Inter-Quartile Range); unit: mg/dL] | 1.04 [0.88 to 1.34] | 1.09 [0.92 to 1.36] | 1.08 [0.9 to 1.35]
Ig levels at entry [Median (Inter-Quartile Range); unit: mg/dL]
  IgG | 699 [560 to 831] | 750 [575 to 923] | 710 [574 to 860]
  IgM | 23 [15 to 47] | 31 [19 to 53] | 29 [17 to 52]
eGFR at entry [Median (Inter-Quartile Range); unit: cc/min/1.73m^2] | 60 [47 to 60] | 60 [50 to 60] | 60 [47 to 60]
Disease status [Count of Participants; unit: Participants]
  Previous relapse | 16 | 17 | 33
  Newly diagnosed | 42 | 40 | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Disease Relapse(s) as Defined by a Birmingham Vasculitis Activity Score for Wegner's Granulomatosis (BVAS/WG) ≥ 2
Description: Relapses recording period was from 6/1/2016 to 12/31/2021. The outcome was reported as the number of participants with disease relapse who had either positive ANCA titers specific for myeloperoxidase (MPO-ANCA) or proteinase 3 (PR3-ANCA). The Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG ) is a form with 34 predefined items grouped into 9 organ systems. The items are clinical features observed in patients with active ANCA vasculitis. Each item has a specified weight of either 3 or 1, depending on whether it reflects major or minor disease activity. The total BVAS/WG score is the weighted sum of individual manifestations that are present and believed to be due to active ANCA vasculitis. Higher scores reflect more active disease. BVAS/WG scores range from 0 to 64.
Time Frame: Median follow-up period of 4.1 years (IQR, 2.5 - 5.0)
Measure: Count of Participants; unit: Participants
Arm/Group | B Cell Reconstitution | Serologic ANCA Flare
Number analyzed (Participants) | 58 | 57
Participants
  PR3 | 1 | 7
  MPO | 4 | 7
Statistical Analysis 1: Comparison: B Cell Reconstitution vs Serologic ANCA Flare; The difference between the two treatment strategies was assessed using the log-rank test. P values of 0.05 were considered significant. Both rows were included and combined in the statistical analysis (ANCA-PR3 and ANCA-MPO) to assess the difference in treatment strategies. Null hypothesis: "No difference in the ANCA and B-cell arm in the probability of relapses"; Test type: Equivalence — Using a two-sided log-rank test with an alpha level of 0.05, a projected relapse risk of 15% in the superior group and 30% in the inferior group, and an estimated enrollment time of 36 months, it was determined that 200 patients were required to detect a significant difference with a power of 0.80. Due to the coronavirus disease 2019 (COVID-19) pandemic and the deleterious impact of rituximab on vaccination efficacy, the trial was concluded before reaching the target enrollment of 200; p = 0.045, Log Rank; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.15 to 0.90]

2. Secondary Outcome: Number of Patients Affected by Serious Adverse Events
Description: Number of patients with serious adverse events (SAEs), including all episodes of late onset neutropenia (LON). SAE are defined in the Serious adverse event section. Serious adverse events were reported over the entire study period (5.5 years)
Time Frame: Median follow-up period of 4.1 years (IQR, 2.5 - 5.0)
Measure: Count of Participants; unit: Participants
Arm/Group | B Cell Reconstitution | Serologic ANCA Flare
Number analyzed (Participants) | 58 | 57
Participants | 15 | 14
Statistical Analysis 1: Comparison: B Cell Reconstitution vs Serologic ANCA Flare; Null hypothesis: "No difference in the proportion of patients with SAEs in each arm"; Test type: Other — chi square test; p = 0.87, Chi-squared

3. Secondary Outcome: Composite of Disease Relapse (Defined a BVAS/WG ≥ 2) and Serious Adverse Events
Description: Number of disease relapse added with the number of SAE in each group
Time Frame: Median follow-up period of 4.1 years (IQR, 2.5 - 5.0)
Measure: Number; unit: Number of events
Arm/Group | B Cell Reconstitution | Serologic ANCA Flare
Number analyzed (Participants) | 58 | 57
Number of events | 27 | 36

4. Secondary Outcome: Number of Patients With Hypogammaglobulinemia
Description: Hypogammaglobulinemia defined as an IgG < 250mg/dL
Time Frame: Median follow-up period of 4.1 years (IQR, 2.5 - 5.0)
Measure: Count of Participants; unit: Participants
Arm/Group | B Cell Reconstitution | Serologic ANCA Flare
Number analyzed (Participants) | 58 | 57
Participants | 1 | 0

5. Secondary Outcome: Patient Survival
Description: number of deaths throughout the study.
Time Frame: 5.5 years
Measure: Number; unit: number of deaths
Arm/Group | B Cell Reconstitution | Serologic ANCA Flare
Number analyzed (Participants) | 58 | 57
number of deaths | 2 | 0

6. Secondary Outcome: Health-related Quality of Life as Assessed by the Short Form Health Survey (SF-36) Scores
Description: The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and is commonly used in health economics as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Assessed throughout the study period, every 6 months unless such time point was not reached or was missed by the patient. Median follow-up period is of 4.1 years (IQR, 2.5 - 5.0)
Population: We collected data using the SF-36 on the quality of life due to its importance in the long-term treatment of ANCA vasculitis. Questionnaires were given to patients every 6 months throughout the study period. Some participants do not have scores at certain time points due to either a missed visit or not being enrolled anymore in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B Cell Reconstitution | Serologic ANCA Flare
Number analyzed (Participants) | 58 | 57
score on a scale
  Physical functioning at 6 months | 84 (19) | 82 (23)
  Role functioning/physical at 6 months | 66 (40) | 65 (45)
  Role functioning/emotional at 6 months | 79 (34) | 75 (41)
  Energy/fatigue at 6 months | 65 (15) | 67 (23)
  Emotional well-being at 6 months | 83 (12) | 81 (16)
  Social functioning at 6 months | 89 (19) | 88 (21)
  Pain at 6 months | 79 (23) | 82 (20)
  General health at 6 months | 66 (15) | 63 (20)
  Physical functioning at 36 months: number analyzed (Participants) | 18 | 18
  Physical functioning at 36 months | 74 (27) | 88 (19)
  Role functioning/physical at 36 months: number analyzed (Participants) | 18 | 18
  Role functioning/physical at 36 months | 50 (47) | 79 (36)
  Role functioning/emotional at 36 months: number analyzed (Participants) | 18 | 18
  Role functioning/emotional at 36 months | 65 (46) | 82 (27)
  Energy/fatigue at 36 months: number analyzed (Participants) | 18 | 18
  Energy/fatigue at 36 months | 58 (17) | 73 (17)
  Emotional well-being at 36 months: number analyzed (Participants) | 18 | 18
  Emotional well-being at 36 months | 76 (19) | 84 (10)
  Social functioning at 36 months: number analyzed (Participants) | 18 | 18
  Social functioning at 36 months | 83 (25) | 95 (13)
  Pain at 36 months: number analyzed (Participants) | 18 | 18
  Pain at 36 months | 69 (23) | 87 (16)
  General health at 36 months: number analyzed (Participants) | 18 | 18
  General health at 36 months | 60 (20) | 70 (20)
  Physical functioning at 12 months: number analyzed (Participants) | 35 | 50
  Physical functioning at 12 months | 79 (24) | 82 (23)
  Role functioning/physical at 12 months: number analyzed (Participants) | 35 | 50
  Role functioning/physical at 12 months | 61 (43) | 63 (43)
  Role functioning/emotional at 12 months: number analyzed (Participants) | 35 | 50
  Role functioning/emotional at 12 months | 82 (34) | 68 (42)
  Energy/ fatigue at 12 months: number analyzed (Participants) | 35 | 50
  Energy/ fatigue at 12 months | 65 (20) | 65 (22)
  Emotional well-being at 12 months: number analyzed (Participants) | 35 | 50
  Emotional well-being at 12 months | 86 (11) | 81 (14)
  Social functioning at 12 months: number analyzed (Participants) | 35 | 50
  Social functioning at 12 months | 92 (18) | 86 (22)
  Pain at 12 months: number analyzed (Participants) | 35 | 50
  Pain at 12 months | 81 (19) | 80 (21)
  General health at 12 months: number analyzed (Participants) | 35 | 50
  General health at 12 months | 66 (17) | 63 (21)
  Physical functioning at 18 months: number analyzed (Participants) | 39 | 40
  Physical functioning at 18 months | 83 (19) | 82 (25)
  Role functioning/physical at 18 months: number analyzed (Participants) | 39 | 40
  Role functioning/physical at 18 months | 70 (41) | 62 (44)
  Role functioning/emotional at 18 months: number analyzed (Participants) | 39 | 40
  Role functioning/emotional at 18 months | 88 (29) | 74 (42)
  Energy/fatigue at 18 months: number analyzed (Participants) | 39 | 40
  Energy/fatigue at 18 months | 69 (14) | 68 (17)
  Emotional well-being at 18 months: number analyzed (Participants) | 39 | 40
  Emotional well-being at 18 months | 85 (9) | 81 (13)
  Social functioning at 18 months: number analyzed (Participants) | 39 | 40
  Social functioning at 18 months | 96 (9) | 92 (16)
  Pain at 18 months: number analyzed (Participants) | 39 | 40
  Pain at 18 months | 84 (18) | 82 (19)
  General health at 18 months: number analyzed (Participants) | 39 | 40
  General health at 18 months | 68 (17) | 67 (18)
  Physical functioning at 24 months: number analyzed (Participants) | 34 | 34
  Physical functioning at 24 months | 83 (24) | 88 (15)
  Role functioning/physical at 24 months: number analyzed (Participants) | 34 | 34
  Role functioning/physical at 24 months | 71 (40) | 71 (42)
  Role functioning/emotional at 24 months: number analyzed (Participants) | 34 | 34
  Role functioning/emotional at 24 months | 84 (33) | 80 (38)
  Energy/fatigue at 24 months: number analyzed (Participants) | 34 | 34
  Energy/fatigue at 24 months | 68 (15) | 76 (13)
  Emotional well-being at 24 months: number analyzed (Participants) | 34 | 34
  Emotional well-being at 24 months | 82 (15) | 85 (12)
  Social functioning at 24 months: number analyzed (Participants) | 34 | 34
  Social functioning at 24 months | 91 (20) | 94 (14)
  Pain at 24 months: number analyzed (Participants) | 34 | 34
  Pain at 24 months | 81 (22) | 82 (15)
  General health at 24 months: number analyzed (Participants) | 34 | 34
  General health at 24 months | 69 (15) | 70 (16)
  Physical functioning at 30 months: number analyzed (Participants) | 21 | 32
  Physical functioning at 30 months | 85 (17) | 88 (17)
  Role functioning/physical at 30 months: number analyzed (Participants) | 21 | 32
  Role functioning/physical at 30 months | 74 (38) | 72 (40)
  Role functioning/emotional at 30 months: number analyzed (Participants) | 21 | 32
  Role functioning/emotional at 30 months | 87 (27) | 80 (39)
  Energy/fatigue at 30 months: number analyzed (Participants) | 21 | 32
  Energy/fatigue at 30 months | 64 (16) | 72 (19)
  Emotional well-being at 30 months: number analyzed (Participants) | 21 | 32
  Emotional well-being at 30 months | 81 (12) | 84 (14)
  Social functioning at 30 months: number analyzed (Participants) | 21 | 32
  Social functioning at 30 months | 90 (19) | 94 (12)
  Pain at 30 months: number analyzed (Participants) | 21 | 32
  Pain at 30 months | 86 (17) | 83 (18)
  General health at 30 months: number analyzed (Participants) | 21 | 32
  General health at 30 months | 60 (14) | 70 (16)
  Physical functioning at 42 months: number analyzed (Participants) | 13 | 15
  Physical functioning at 42 months | 76 (25) | 82 (24)
  Role functioning/physical at 42 months: number analyzed (Participants) | 13 | 15
  Role functioning/physical at 42 months | 58 (49) | 60 (40)
  Role functioning/emotional at 42 months: number analyzed (Participants) | 13 | 15
  Role functioning/emotional at 42 months | 67 (47) | 76 (37)
  Energy/fatigue at 42 months: number analyzed (Participants) | 13 | 15
  Energy/fatigue at 42 months | 60 (19) | 70 (24)
  Emotional well-being at 42 months: number analyzed (Participants) | 13 | 15
  Emotional well-being at 42 months | 77 (18) | 85 (12)
  Social functioning at 42 months: number analyzed (Participants) | 13 | 15
  Social functioning at 42 months | 85 (15) | 87 (24)
  Pain at 42 months: number analyzed (Participants) | 13 | 15
  Pain at 42 months | 83 (16) | 82 (21)
  General health at 42 months: number analyzed (Participants) | 13 | 15
  General health at 42 months | 59 (13) | 63 (22)
  Physical functioning at 48 months: number analyzed (Participants) | 6 | 1
  Physical functioning at 48 months | 65 (29) | 95 (0)
  Role functioning/physical at 48 months: number analyzed (Participants) | 6 | 1
  Role functioning/physical at 48 months | 67 (52) | 100 (0)
  Role functioning/emotional at 48 months: number analyzed (Participants) | 6 | 1
  Role functioning/emotional at 48 months | 67 (52) | 100 (0)
  Energy/fatigue at 48 months: number analyzed (Participants) | 6 | 1
  Energy/fatigue at 48 months | 52 (21) | 75 (0)
  Emotional well-being at 48 months: number analyzed (Participants) | 6 | 1
  Emotional well-being at 48 months | 73 (29) | 85 (0)
  Social functioning at 48 months: number analyzed (Participants) | 6 | 1
  Social functioning at 48 months | 65 (41) | 100 (0)
  Pain at 48 months: number analyzed (Participants) | 6 | 1
  Pain at 48 months | 70 (32) | 80 (0)
  General health at 48 months: number analyzed (Participants) | 6 | 1
  General health at 48 months | 61 (22) | 75 (0)
  Physical functioning at 54 months: number analyzed (Participants) | 4 | 0
  Physical functioning at 54 months | 88 (14) |
  Role functioning/physical at 54 months: number analyzed (Participants) | 4 | 0
  Role functioning/physical at 54 months | 50 (58) |
  Role functioning/emotional at 54 months: number analyzed (Participants) | 4 | 0
  Role functioning/emotional at 54 months | 67 (38) |
  Energy/fatigue at 54 months: number analyzed (Participants) | 4 | 0
  Energy/fatigue at 54 months | 67 (19) |
  Emotional well-being at 54 months: number analyzed (Participants) | 4 | 0
  Emotional well-being at 54 months | 84 (5) |
  Social functioning at 54 months: number analyzed (Participants) | 4 | 0
  Social functioning at 54 months | 84 (19) |
  Pain at 54 months: number analyzed (Participants) | 4 | 0
  Pain at 54 months | 81 (26) |
  General health at 54 months: number analyzed (Participants) | 4 | 0
  General health at 54 months | 59 (6) |
  Physical functioning at 60 months: number analyzed (Participants) | 3 | 3
  Physical functioning at 60 months | 72 (25) | 92 (3)
  Role functioning/physical at 60 months: number analyzed (Participants) | 3 | 3
  Role functioning/physical at 60 months | 33 (58) | 100 (0)
  Role functioning/emotional at 60 months: number analyzed (Participants) | 3 | 3
  Role functioning/emotional at 60 months | 100 (0) | 89 (19)
  Energy/fatigue at 60 months: number analyzed (Participants) | 3 | 3
  Energy/fatigue at 60 months | 48 (24) | 71 (14)
  Emotional well-being at 60 months: number analyzed (Participants) | 3 | 3
  Emotional well-being at 60 months | 82 (10) | 83 (6)
  Social functioning at 60 months: number analyzed (Participants) | 3 | 3
  Social functioning at 60 months | 63 (38) | 92 (14)
  Pain at 60 months: number analyzed (Participants) | 3 | 3
  Pain at 60 months | 53 (13) | 83 (13)
  General health at 60 months: number analyzed (Participants) | 3 | 3
  General health at 60 months | 58 (32) | 70 (23)

7. Secondary Outcome: Mean Number of Rituximab Infusions Per Subject
Description: The rituximab utilization was measured in how many times a subject received Rituximab throughout the study which was then averaged for all subjects in each treatment arm, including those who did not receive any infusion.
Time Frame: Median follow-up period of 4.1 years (IQR, 2.5 - 5.0)
Measure: Mean (Standard Deviation); unit: Infusions per subject
Arm/Group | B Cell Reconstitution | Serologic ANCA Flare
Number analyzed (Participants) | 58 | 57
Infusions per subject | 3.6 (2.4) | 0.5 (1.5)
Statistical Analysis 1: Comparison: B Cell Reconstitution vs Serologic ANCA Flare; Null hypothesis: no difference in the mean number of infusions per patient in each arm; Test type: Other; p < 0001, t-test, 2 sided

8. Secondary Outcome: Organ Damage as Assessed by the Vasculitis Damage Index (VDI).
Description: The Vasculitis Damage Index (VDI) is a validated formal assessment tool in ANCA-associated vasculitis clinical trials. The VDI distinguishes vasculitis-induced chronic damage from active inflammation or persistent disease. Each item represents a disease manifestation and is given a score (of 1) if present for at least 3 months. Neither the cause of damage (vasculitis vs treatment) nor an ongoing activity are taken into consideration. The VDI includes 64 items categorized into 11 groups (by organ system) and the scored items are summed to give a total score ranging from 0 to 64. A higher score means more accrued damage.
Time Frame: 3 years starting at inclusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B Cell Reconstitution | Serologic ANCA Flare
Number analyzed (Participants) | 58 | 57
score on a scale
  VDI at inclusion | 1.27 (1.24) | 1.07 (1.11)
  VDI at 3 years | 1.42 (1.11) | 1.08 (1.16)
Statistical Analysis 1: Comparison: B Cell Reconstitution vs Serologic ANCA Flare; Null hypothesis: there is no difference in the mean change from baseline Vasculitis Damage Index between each arm. A t-test was used; Test type: Other; p = 0.17, t-test, 2 sided; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.34 to -0.06]

9. Secondary Outcome: Number of Major Relapses Defined as a BVAS/WG ≥ 3
Description: The Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG ) is a form with 34 predefined items grouped into 9 organ systems. The items are clinical features observed in patients with active ANCA vasculitis. Each item has a specified weight of either 3 or 1, depending on whether it reflects major or minor disease activity. The total BVAS/WG score is the weighted sum of individual manifestations that are present and believed to be due to active ANCA vasculitis. Higher scores reflect more active disease. BVAS/WG scores range from 0 to 64.
Time Frame: Median follow-up period of 4.1 years (IQR, 2.5 - 5.0)
Measure: Number; unit: number of events
Arm/Group | B Cell Reconstitution | Serologic ANCA Flare
Number analyzed (Participants) | 58 | 57
number of events | 4 | 7
Statistical Analysis 1: Comparison: B Cell Reconstitution vs Serologic ANCA Flare; The difference between the two treatment strategies was assessed using the log-rank test. P values of 0.05 were considered significant. Null hypothesis: "No difference in the ANCA and B-cell arm in the probability of relapses"; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.42, Log Rank; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [0.50 to 5.36]

10. Secondary Outcome: Number of Infections
Description: Number of infections mild and severe, whether they were treated or not with antibiotics
Time Frame: Median follow-up period of 4.1 years (IQR, 2.5 - 5.0)
Measure: Number; unit: number of events
Arm/Group | B Cell Reconstitution | Serologic ANCA Flare
Number analyzed (Participants) | 58 | 57
number of events
  Serious Adverse Events- Infections | 12 | 6
  Adverse Events- Infections | 72 | 59

ADVERSE EVENTS:
Time Frame: June 1 2016 to December 2021 (5 years and 6 months). The earliest Adverse event reported was on 2/6/2017 and the latest adverse event reported was on 12/25/2021
Description: All adverse events will be reported per PHRC guidelines which includes unanticipated problems involving risks to subjects/others, including adverse events, within 5 working days/7 calendar days of the date that the investigator first became aware of the problem.
Arm/Group | B Cell Reconstitution | Serologic ANCA Flare
All-Cause Mortality (participants affected / at risk) | 2/58 | 0/57
Serious Adverse Events (participants affected / at risk) | 15/58 | 14/57
Other Adverse Events (participants affected / at risk) | 46/58 | 44/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B Cell Reconstitution (N=58) | Serologic ANCA Flare (N=57)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Urinary Track Infection (Infections and infestations) | 1 (1) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 6 (6) | 1 (1)
Cancer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Squamous cell carcinoma
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Thromboembolic disease
Neutropenia (Immune system disorders) | 1 (1) | 0 (0)
Death (Infections and infestations) | 2 (2) | 0 (0) — all were due to COVID-19
Psychiatric Disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Transient ischemic attacks (Vascular disorders) | 0 (0) | 1 (1)
Urinary retention and elevated creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)
Rectal bleeding status post colonoscopy (Gastrointestinal disorders) | 0 (0) | 1 (1)
bleeding gastric nodule (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asymptomatic AKI (Renal and urinary disorders) | 0 (0) | 1 (1) — Cr to 1.9 from baseline 1.5. Kidney biopsy 10/22/19 showed chronic active interstitial nephritis
Gallstone pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pulmonary edema in setting of fluid resuscitation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lumbar disc herniation, cervical and lumbar stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Renal Calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
New elevated IgM in setting of longstanding pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain, LAD stenosis and RAD stenosis (Cardiac disorders) | 0 (0) | 1 (1) — Admitted with chest pain - arteriogram at cath lab found LAD: 99% mid LAD stenosis; RCA: 95% stenosis with an early branching acute marginal.
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease- Three-vessel disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis and Heart failure with preserved ejection fraction (Cardiac disorders) | 1 (1) | 0 (0) — Myocarditis was the first diagnosis. New diagnosis of HFpEF later on.
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B Cell Reconstitution (N=58) | Serologic ANCA Flare (N=57)
Upper Respiratory Infection (Cold) (Infections and infestations) | 21 (28) | 17 (24) — Cold, pharyngitis and other URI. Sinusitis are not included if isolated and specified in the description of event.
Urinary Track Infection (Renal and urinary disorders) | 5 (9) | 6 (7)
Gout flare (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 8 (9)
Sinusitis (Infections and infestations) | 3 (5) | 7 (8)
COVID-19 Positive (Infections and infestations) | 9 (9) | 4 (4)
Allergic Reaction to Rituximab Infusion (Immune system disorders) | 3 (3) | 1 (1)
Allergic reaction unrelated to Rituximab (Immune system disorders) | 1 (1) | 0 (0)
Vaginitis (Infections and infestations) | 1 (1) | 2 (2) — One due to yeasts, for the two other the cause is unknown
Asymptomatic Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Right thigh pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Mild, not injury related, for 2 days and resolved.
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Heart murmurs (Cardiac disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
pleural infection (Infections and infestations) | 0 (0) | 1 (1)
Myalgias and arthralgias. Severe pains and frank arthritis in knees. (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pleuritic chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — CTA scan negative for PE but positive for pleural inflammatory process
Mild fatty replacement of the liver (Hepatobiliary disorders) | 1 (1) | 0 (0)
Metacarpophalangeal tenderness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Right 1st MCP
Headache/ Migraine (Nervous system disorders) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 4 (5)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Conduction disorder (LBBB) (Cardiac disorders) | 0 (0) | 1 (1)
Fall injury (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) — * Hip and back pain * thumb fracture and hit head without LOC, headaches or confusion * shoulder injury
colonoscopy finding:tubulovillous adenomatous colon poplyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Rash in distribution of trigeminal nerve - consistent with zoster (Infections and infestations) | 1 (1) | 0 (0)
Hypotension, fatigue, cough, HA, fever, malaise, volume depletion from high dose valtrex reaction (General disorders) | 1 (1) | 0 (0)
Urine cx positive for E.coli (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 2 (2)
Paronychia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Elevated Liver Function Tests (Hepatobiliary disorders) | 0 (0) | 3 (3) — LFTs for each patients: * ALT 144. AST 82. Patient stopped taking supplement * ALT 62. Resolved at next visit * ALT 225, AST 192, Alk-Phos 174
Mandibular pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neutropenia (Immune system disorders) | 1 (1) | 1 (1)
Epistaxis (Vascular disorders) | 1 (1) | 1 (1)
Jaw swelling, (Immune system disorders) | 1 (1) | 0 (0) — internal swelling and sensation of fullness in jaw. Related AE, led to stop cephalexin.
Distal Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — New edema and clot in lower leg near ankle
Stomach discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) — Stomach discomfort. Mild ache and cramping pain over last month. Patient noted start coincided with switch to amlodipine
Sore throat (Infections and infestations) | 1 (1) | 0 (0) — sore throat; symptoms consistent of swollen lymph node, likely secondary viral or bacterial infection.
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) — Non serious and moderate
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
RLL possibe airspace disease and/or atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Degenerative disk disease of c-spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertigo (General disorders) | 1 (1) | 0 (0)
Diarrhea (Infections and infestations) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Lung opacity and nodule (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Dizziness (Investigations) | 1 (1) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 2 (2)
Leg Edema (Cardiac disorders) | 1 (1) | 1 (1)
Ear pain (Infections and infestations) | 1 (1) | 1 (1) — Possibly due to infection
Surgical procedure (Surgical and medical procedures) | 1 (1) | 1 (2)
Tooth infection (Infections and infestations) | 2 (2) | 0 (0)
Skin rash on arms and legs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Raised red rash on bilateral arms and legs. Not itchy or painful. Lesions come and go
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) — Annual ECG with new atrial flutter. Patient asymptomatic
Achilles tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Bilateral Achilles tendon pain. Patient had taken levaquin ~1 month prior
Shoulder cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Shoulder cyst. Now large and tense
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Atrial fibrillation Mild
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exertional dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Exertional dyspnea. Requires break after 1-2 blocks; a/w diaphoresis. DDx includes poorly controlled asthma vs deconditioning vs coronary disease
Prostatic Obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Herpes simplex virus rash (Infections and infestations) | 1 (1) | 0 (0) — Herpes simplex virus. Vesicular rash on lower lip and chin. Mostly on left and on midline
Heart palpitations (Cardiac disorders) | 0 (0) | 1 (1) — 3x/week for 3 weeks lasting less than 1 min. No pain, SOB or numbness.
Adrenal incidentaloma (Endocrine disorders) | 0 (0) | 1 (1)
Conduction disorder- Non-specific intraventricular block (Cardiac disorders) | 0 (0) | 1 (1) — Non-specific intraventricular block (conduction disorder). QRS 128ms.
Bilateral impacted cerumen (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Herpes simplex cold sore (Infections and infestations) | 1 (1) | 0 (0) — Cold sore on lip, treated with valtrex
Balanitis (Infections and infestations) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ankle soreness and swelling post exercize (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Left ankle soreness with severe swelling after walking a lot in France
Bilateral swelling in the ankle and high blood pressure (Immune system disorders) | 0 (0) | 1 (1)
Knee arthritis (Immune system disorders) | 1 (1) | 0 (0) — New left acute knee arthritis. Initially thought consistent with gout, but patient on uloric for past 2 years. Uric acid 5.5
Esophageal narrowing (Gastrointestinal disorders) | 0 (0) | 1 (1)
Recurrent Lightheadedness (Vascular disorders) | 0 (0) | 1 (1) — Patient experienced recurrent lightheadedness after increasing Losartan HCT from 50/12.5 to 100/25.
Cardiac arrythmia (Cardiac disorders) | 0 (0) | 1 (1)
Sores in mouth (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Sores in mouth attributed to Invisalign
Infection lower eye lid (Infections and infestations) | 1 (1) | 0 (0) — Treated with polymyxin drops
Polyarticular arthritis (Immune system disorders) | 0 (0) | 1 (1) — Developed large toe arthritis then wrist, finger, ankle swelling.
Infection on left side of the face (Infections and infestations) | 1 (1) | 0 (0) — Non serious, related and treated with 5 days of antibiotics.
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — epigastric pain radiating to back and RUQ. Associated with nausea and 3 episodes emesis
Eye and face swelling (Infections and infestations) | 0 (0) | 1 (1) — Present to the ED with right eye swelling and pain. Right chin swelling and pain. Subject was prescribed doxycycline cyclate 100mg tablet
Arm, shoulder and neck pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — On and off, for 10 minutes. Not associated with exertion.
Shingles (Infections and infestations) | 1 (1) | 0 (0) — Shingles. C4 distribution. Right
Syncopal episode (Cardiac disorders) | 0 (0) | 1 (1)
Rash on chest - Allergy (Immune system disorders) | 1 (1) | 0 (0) — Rash on chest for 5 days. Pt believes caused by perfume or lotion
Scleritis (Infections and infestations) | 0 (0) | 1 (1) — Medial right eye scleritis treated emergently with prednisolone x 2 weeks, with improvement over 24 hours and no return of symptoms after drops stopped. Presented with gritty feeling whe blinking. Attributed to foreign body in eye

LIMITATIONS AND CAVEATS:
The trial has several limitations:

1. It was open-label.
2. it only enrolled patients on continuous B cell depletion for a minimum of 2 years
3. it took place in a single center.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT02749292/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT02749292/ICF_001.pdf